CLINICAL TRIAL: NCT00358748
Title: Early Use of Hydrocortisone in Hypotensive Very Low Birth Weight Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Research Inc. (Industry)
Responsible Party: Dr. Horacio Osiovich, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C05-0006
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Neonatal Hypotension
Keywords: Preterm; hypotension; steroids; hydrocortisone
MeSH Terms: conditions — Premature Birth; Hypotension | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydrocortisone — See detailed description above.

SUMMARY:
The purpose of this study is to investigate the early use of hydrocortisone in hypotensive very low birth weight infants.

Based on the observations that:

* hypotension is a common problem in very low birthweight infants and is associated with brain injury and poor neurological outcomes;
* some infants are refractory to standard treatment (volume expansion and vasopressors), which is not exempt of adverse effects;
* relative adrenal insufficiency has been described in this population; we hypothesize that hydrocortisone is effective in the treatment of hypotension in this population and reduce the need for vasopressors.

DETAILED DESCRIPTION:
Eligible infants will be randomly assigned to receive hydrocortisone or placebo, using sequentially numbered, preassigned treatment designations in sealed, opaque envelopes. The study drug will be randomly assigned to each patient number, in advance, using a computer-based random number generator.

Hydrocortisone and placebo doses will be prepared and provided by the hospital pharmacy following the assigned study number. Active and placebo drug solutions will be completely indistinguishable.

Infants of multiple gestations will be randomized as separate subjects. Crossover between study groups is not allowed. Physicians involved in the care of the infants will be blinded to treatment group allocation.

If the infant remains hypotensive after a Normal Saline (NS) bolus 10 ml/kg, blood for serum cortisol level determination will be drawn and hydrocortisone or an equivalent volume of NS placebo will be administered intravenously as follows: first dose immediately after randomization 2 mg/kg; 6 hours after 1 mg/kg q6h for 3 doses; followed by 0.5 mg/kg q6hs for 4 doses. If an infant responds to the initial dose of NS but becomes hypotensive within 1 hour after will also be randomized, otherwise another NS bolus could be administered.

Initiation and escalation of inotropes:

Concurrently with the first dose of study drug, dopamine infusion will be started at 5 mcg/kg/minute, increasing stepwise to a maximum of 15 mcg/kg/minute. If hypotension persists an epinephrine infusion at 0.05 mcg/kg/min will be added and increased stepwise if necessary. The aim is to maintain mean blood pressure (MBP) above the hypotensive limit defined in the inclusion criteria.

Weaning of inotropes:

Once normotension has been maintained for 1 hour or MBP > 40 mmHg for 15 minutes, weaning should be started. Dopamine infusion will be reduced first, as tolerated, to 5 mcg/kg/minute. If the subject is on epinephrine infusion the dose will be reduced stepwise to 0.05 mcg/kg/minute and discontinued. When the subject is off epinephrine and/or dopamine at 5 mcg/kg/minute, dopamine will be discontinued. If at any time hypotension recurs, weaning should be held and increased inotropes dose as per escalation algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 30 weeks, Birth weight ≤ 1250 grams and ≤ 48 hours age;
* Umbilical or peripheral arterial catheter in place;
* Invasive mean blood pressure < gestational age in completed weeks after 1 Normal Saline bolus 10 ml/kg;
* Parental/legal guardian consent.

Exclusion Criteria:

* Clear evidence of hypovolemia (blood loss);
* Chromosomal abnormalities;
* Hydrops fetalis;
* Major congenital anomalies;
* Cardiac lesions other than patent ductus arteriosus.

Ages: 48 Hours to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Total cumulative dose of dopamine at 48 hours of study drug administration and by day 7 of life | 7 days

SECONDARY OUTCOMES:
Total cumulative dose of epinephrine and total dose of fluids at 48 hours of study drug administration and by day 7 of life | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Osiovich, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Division of Neonatology, Children's and Women's Health Centre, Vancouver, British Columbia, Canada